CLINICAL TRIAL: NCT01621711
Title: Continuing Care Following Drug Abuse Treatment: Linkage With Primary Care
Acronym: Linkage
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Kaiser Foundation Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-01606
Record Dates: First submitted 2012-06-11; First posted 2012-06-18 (Estimated); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Substance Abuse; Substance Dependence; Substance, Addiction; Alcohol Abuse
Keywords: substance abuse; Substance Dependence; Substance, addiction; Alcohol Abuse; prevention and control; preventative health services; patient centered care
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Usual CD treatment, including therapy groups and individual counseling sessions, and six 45-min medical education groups. Physician appointments, pharmacotherapy, and SUD medications were be available as needed.
- Linkage patient activation intervention (Experimental): Usual Care with the exception that the six 45-min Linkage patient activation education groups replaced the six 45-min Usual Care medical education groups, plus a linkage phone call (and/or a facilitated email) with the patient, clinician, and Primary Care physician.
  Interventions: Behavioral: Linkage patient activation intervention

INTERVENTIONS:
Behavioral: Linkage patient activation intervention — Usual Care plus Linkage encompassed Usual Care with the exception that the six 45-min Linkage patient activation education groups replaced the six 45-min Usual Care medical education groups, plus a linkage phone call (and/or a facilitated email) with the patient, clinician, and Primary Care physician.
  The patient activation intervention components -- 1) six 45-min Linkage sessions on activation regarding overall health behaviors and 2) a linkage phone call (and/or a facilitated email) with the patient, clinician, and PC physician -- were delivered by a clinical psychologist.
  Arms: Linkage patient activation intervention

SUMMARY:
This component of a larger Center of Research Excellence Grant improves treatment for drug abuse by developing effective linkages between specialty drug treatment and primary health care.

DETAILED DESCRIPTION:
This is a longitudinal two-arm quasi-experimental 3-month alternating off/on design over a 30 month period in which, after a random start, the Linkage condition alternately is added to Usual Care in the Chemical Dependency (CD) clinic and then removed. We compare Usual Care to Usual Care plus Linkage. Follow-up interviews will be conducted at 6, 12 and 24 months. The Linkage intervention includes Usual Care plus 1) sessions on activation regarding overall health behaviors and on selecting a Primary Care physician and communicating with him/her, and 2) a linkage phone call (and/or a facilitated email) with the patient, clinician, and Primary Care physician. The intervention aims to place drug abuse problems in the context of overall health and health care and to activate patients to increase involvement in their own health care.

ELIGIBILITY:
Inclusion Criteria:

* Research participants will be adult patients at the Kaiser Permanente San Francisco Chemical Dependency Recovery Program, who have completed 2 weeks of treatment.

Exclusion Criteria:

* Patients with a diagnosis of dementia, mental retardation, or who are actively psychotic or suicidal will be excluded by their clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2011-03; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
patient activation measure | 6 months post baseline
  Measured by Patient Activation Measure (PAM) from interview data
patient engagement in health care (including patient portal use, familiarity and satisfaction with Primary Care physician, and CD treatment length of stay) | 6 months post baseline
  Measured by data from interviews and Electronic Health Record (EHR)
Substance use and mental health outcomes | 6 months post baseline
  Measures include past 30-day alcohol, drug and total abstinence; Patient Health Questionnaire (PHQ-9) and Addiction Severity Index using interview data

SECONDARY OUTCOMES:
patient activation measure at 12 and 24 months | 12 and 24 months post baseline
  Measured by Patient Activation Measure (PAM) from interview data
patient engagement in health care at 12 and 24 months | 12 and 24 months post baseline
  Measured by data from interviews and Electronic Health Record (EHR)
Substance use and mental health outcomes at 12 and 24 months | 12 and 24 months post baseline
  Measures include past 30-day alcohol, drug and total abstinence; Patient Health Questionnaire (PHQ-9) and Addiction Severity Index using interview data
Health care utilization and cost | 12 and 24 months post baseline
  Measured by data from interviews and adminstrative data

CONTACTS AND LOCATIONS:
Overall Officials: Constance M Weisner, DrPH, LCSW, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Chemical Dependency Recovery Program, San Francisco, California, United States

REFERENCES:
- [Background] Saitz R, Horton NJ, Larson MJ, Winter M, Samet JH. Primary medical care and reductions in addiction severity: a prospective cohort study. Addiction. 2005 Jan;100(1):70-8. doi: 10.1111/j.1360-0443.2005.00916.x. PMID 15598194
- [Background] Mertens JR, Flisher AJ, Satre DD, Weisner CM. The role of medical conditions and primary care services in 5-year substance use outcomes among chemical dependency treatment patients. Drug Alcohol Depend. 2008 Nov 1;98(1-2):45-53. doi: 10.1016/j.drugalcdep.2008.04.007. Epub 2008 Jun 20. PMID 18571875
- [Background] Von Korff M, Gruman J, Schaefer J, Curry SJ, Wagner EH. Collaborative management of chronic illness. Ann Intern Med. 1997 Dec 15;127(12):1097-102. doi: 10.7326/0003-4819-127-12-199712150-00008. PMID 9412313
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness. JAMA. 2002 Oct 9;288(14):1775-9. doi: 10.1001/jama.288.14.1775. PMID 12365965
- [Background] Tsuang MT, Lyons MJ, Eisen SA, Goldberg J, True W, Lin N, Meyer JM, Toomey R, Faraone SV, Eaves L. Genetic influences on DSM-III-R drug abuse and dependence: a study of 3,372 twin pairs. Am J Med Genet. 1996 Sep 20;67(5):473-7. doi: 10.1002/(SICI)1096-8628(19960920)67:53.0.CO;2-L. PMID 8886164
- [Background] Schuckit MA, Smith TL. An 8-year follow-up of 450 sons of alcoholic and control subjects. Arch Gen Psychiatry. 1996 Mar;53(3):202-10. doi: 10.1001/archpsyc.1996.01830030020005. PMID 8611056
- [Background] Dennis M, Scott CK. Managing addiction as a chronic condition. Addict Sci Clin Pract. 2007 Dec;4(1):45-55. doi: 10.1151/ascp074145. PMID 18292710
- [Background] Dennis ML, Scott CK, Funk R, Foss MA. The duration and correlates of addiction and treatment careers. J Subst Abuse Treat. 2005;28 Suppl 1:S51-62. doi: 10.1016/j.jsat.2004.10.013. PMID 15797639
- [Background] Weisner C, Ray GT, Mertens JR, Satre DD, Moore C. Short-term alcohol and drug treatment outcomes predict long-term outcome. Drug Alcohol Depend. 2003 Sep 10;71(3):281-94. doi: 10.1016/s0376-8716(03)00167-4. PMID 12957346
- [Background] Hser YI, Anglin MD, Grella C, Longshore D, Prendergast ML. Drug treatment careers. A conceptual framework and existing research findings. J Subst Abuse Treat. 1997 Nov-Dec;14(6):543-58. doi: 10.1016/s0740-5472(97)00016-0. PMID 9437626
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness: the chronic care model, Part 2. JAMA. 2002 Oct 16;288(15):1909-14. doi: 10.1001/jama.288.15.1909. PMID 12377092
- [Background] Mosen DM, Schmittdiel J, Hibbard J, Sobel D, Remmers C, Bellows J. Is patient activation associated with outcomes of care for adults with chronic conditions? J Ambul Care Manage. 2007 Jan-Mar;30(1):21-9. doi: 10.1097/00004479-200701000-00005. PMID 17170635
- [Background] Schmittdiel J, Mosen DM, Glasgow RE, Hibbard J, Remmers C, Bellows J. Patient Assessment of Chronic Illness Care (PACIC) and improved patient-centered outcomes for chronic conditions. J Gen Intern Med. 2008 Jan;23(1):77-80. doi: 10.1007/s11606-007-0452-5. Epub 2007 Nov 21. PMID 18030539
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Holman H, Lorig K. Patients as partners in managing chronic disease. Partnership is a prerequisite for effective and efficient health care. BMJ. 2000 Feb 26;320(7234):526-7. doi: 10.1136/bmj.320.7234.526. No abstract available. PMID 10688539
- [Background] Wagner EH, Austin BT, Von Korff M. Improving outcomes in chronic illness. Manag Care Q. 1996 Spring;4(2):12-25. PMID 10157259
- [Background] McKay JR, Carise D, Dennis ML, Dupont R, Humphreys K, Kemp J, Reynolds D, White W, Armstrong R, Chalk M, Haberle B, McLellan T, O'Connor G, Pakull B, Schwartzlose J. Extending the benefits of addiction treatment: practical strategies for continuing care and recovery. J Subst Abuse Treat. 2009 Mar;36(2):127-30. doi: 10.1016/j.jsat.2008.10.005. No abstract available. PMID 19161893
- [Background] McKay JR. Continuing care research: what we have learned and where we are going. J Subst Abuse Treat. 2009 Mar;36(2):131-45. doi: 10.1016/j.jsat.2008.10.004. PMID 19161894
- [Background] McKay JR, Carise D. State of the science: Extending the benefits of addiction treatment. J Subst Abuse Treat. 2009 Mar;36(2):172-3. doi: 10.1016/j.jsat.2008.10.007. No abstract available. PMID 19161897
- [Background] McKay JR. Is there a case for extended interventions for alcohol and drug use disorders? Addiction. 2005 Nov;100(11):1594-610. doi: 10.1111/j.1360-0443.2005.01208.x. PMID 16277622
- [Background] McKay JR, Lynch KG, Shepard DS, Pettinati HM. The effectiveness of telephone-based continuing care for alcohol and cocaine dependence: 24-month outcomes. Arch Gen Psychiatry. 2005 Feb;62(2):199-207. doi: 10.1001/archpsyc.62.2.199. PMID 15699297
- [Background] Grella CE, Greenwell L. Treatment needs and completion of community-based aftercare among substance-abusing women offenders. Womens Health Issues. 2007 Jul-Aug;17(4):244-55. doi: 10.1016/j.whi.2006.11.005. Epub 2007 Jun 4. PMID 17544296
- [Background] Godley SH, Godley MD, Wright KL, Funk RR, Petry NM. Contingent reinforcement of personal goal activities for adolescents with substance use disorders during post-residential continuing care. Am J Addict. 2008 Jul-Aug;17(4):278-86. doi: 10.1080/10550490802138798. PMID 18612882
- [Background] Godley MD, Godley SH, Dennis ML, Funk R, Passetti LL. Preliminary outcomes from the assertive continuing care experiment for adolescents discharged from residential treatment. J Subst Abuse Treat. 2002 Jul;23(1):21-32. doi: 10.1016/s0740-5472(02)00230-1. PMID 12127465
- [Background] Godley MD, Godley SH, Dennis ML, Funk RR, Passetti LL. The effect of assertive continuing care on continuing care linkage, adherence and abstinence following residential treatment for adolescents with substance use disorders. Addiction. 2007 Jan;102(1):81-93. doi: 10.1111/j.1360-0443.2006.01648.x. PMID 17207126
- [Background] Ritsher JB, McKellar JD, Finney JW, Otilingam PG, Moos RH. Psychiatric comorbidity, continuing care and mutual help as predictors of five-year remission from substance use disorders. J Stud Alcohol. 2002 Nov;63(6):709-15. doi: 10.15288/jsa.2002.63.709. PMID 12529071
- [Background] Weisner C, Mertens J, Parthasarathy S, Moore C, Lu Y. Integrating primary medical care with addiction treatment: a randomized controlled trial. JAMA. 2001 Oct 10;286(14):1715-23. doi: 10.1001/jama.286.14.1715. PMID 11594896
- [Background] Friedmann PD, Saitz R, Samet JH. Management of adults recovering from alcohol or other drug problems: relapse prevention in primary care. JAMA. 1998 Apr 15;279(15):1227-31. doi: 10.1001/jama.279.15.1227. PMID 9555766
- [Background] Friedmann PD, Hendrickson JC, Gerstein DR, Zhang Z, Stein MD. Do mechanisms that link addiction treatment patients to primary care influence subsequent utilization of emergency and hospital care? Med Care. 2006 Jan;44(1):8-15. doi: 10.1097/01.mlr.0000188913.50489.77. PMID 16365607
- [Background] Friedmann PD, Zhang Z, Hendrickson J, Stein MD, Gerstein DR. Effect of primary medical care on addiction and medical severity in substance abuse treatment programs. J Gen Intern Med. 2003 Jan;18(1):1-8. doi: 10.1046/j.1525-1497.2003.10601.x. PMID 12534757
- [Background] McLellan AT, Alterman AI, Metzger DS, Grissom GR, Woody GE, Luborsky L, O'Brien CP. Similarity of outcome predictors across opiate, cocaine, and alcohol treatments: role of treatment services. J Consult Clin Psychol. 1994 Dec;62(6):1141-58. doi: 10.1037//0022-006x.62.6.1141. PMID 7860812
- [Background] Umbricht-Schneiter A, Ginn DH, Pabst KM, Bigelow GE. Providing medical care to methadone clinic patients: referral vs on-site care. Am J Public Health. 1994 Feb;84(2):207-10. doi: 10.2105/ajph.84.2.207. PMID 8296941
- [Background] Samet JH, Larson MJ, Horton NJ, Doyle K, Winter M, Saitz R. Linking alcohol- and drug-dependent adults to primary medical care: a randomized controlled trial of a multi-disciplinary health intervention in a detoxification unit. Addiction. 2003 Apr;98(4):509-16. doi: 10.1046/j.1360-0443.2003.00328.x. PMID 12653820
- [Background] Saitz R, Larson MJ, Horton NJ, Winter M, Samet JH. Linkage with primary medical care in a prospective cohort of adults with addictions in inpatient detoxification: room for improvement. Health Serv Res. 2004 Jun;39(3):587-606. doi: 10.1111/j.1475-6773.2004.00246.x. PMID 15149480
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Background] Stein MD. Medical consequences of substance abuse. Psychiatr Clin North Am. 1999 Jun;22(2):351-70. doi: 10.1016/s0193-953x(05)70081-2. PMID 10385938
- [Background] Mertens JR, Lu YW, Parthasarathy S, Moore C, Weisner CM. Medical and psychiatric conditions of alcohol and drug treatment patients in an HMO: comparison with matched controls. Arch Intern Med. 2003 Nov 10;163(20):2511-7. doi: 10.1001/archinte.163.20.2511. PMID 14609789
- [Background] Chou SP, Grant BF, Dawson DA. Medical consequences of alcohol consumption--United States, 1992. Alcohol Clin Exp Res. 1996 Nov;20(8):1423-9. doi: 10.1111/j.1530-0277.1996.tb01144.x. PMID 8947320
- [Background] Redelmeier DA, Tan SH, Booth GL. The treatment of unrelated disorders in patients with chronic medical diseases. N Engl J Med. 1998 May 21;338(21):1516-20. doi: 10.1056/NEJM199805213382106. PMID 9593791
- [Background] Gonzales JJ, Insel TR. The conundrum of co-occurring mental and substance use disorders: opportunities for research. Biol Psychiatry. 2004 Nov 15;56(10):723-5. doi: 10.1016/j.biopsych.2004.09.007. No abstract available. PMID 15556114
- [Background] Volkow ND. The reality of comorbidity: depression and drug abuse. Biol Psychiatry. 2004 Nov 15;56(10):714-7. doi: 10.1016/j.biopsych.2004.07.007. No abstract available. PMID 15556111
- [Background] Montoya ID. Infectious diseases and anemia in a sample of out-of-treatment drug users. Am J Manag Care. 1998 Sep;4(9):1257-64. PMID 10185976
- [Background] Moos RH, Brennan PL, Mertens JR. Diagnostic subgroups and predictors of one-year re-admission among late-middle-aged and older substance abuse patients. J Stud Alcohol. 1994 Mar;55(2):173-83. doi: 10.15288/jsa.1994.55.173. PMID 8189738
- [Background] Bobo JK, Lando HA, Walker RD, McIlvain HE. Predictors of tobacco quit attempts among recovering alcoholics. J Subst Abuse. 1996;8(4):431-43. doi: 10.1016/s0899-3289(96)90004-8. PMID 9058355
- [Background] Compton WM, Thomas YF, Stinson FS, Grant BF. Prevalence, correlates, disability, and comorbidity of DSM-IV drug abuse and dependence in the United States: results from the national epidemiologic survey on alcohol and related conditions. Arch Gen Psychiatry. 2007 May;64(5):566-76. doi: 10.1001/archpsyc.64.5.566. PMID 17485608
- [Background] Kalman D. Smoking cessation treatment for substance misusers in early recovery: a review of the literature and recommendations for practice. Subst Use Misuse. 1998 Aug;33(10):2021-47. doi: 10.3109/10826089809069815. PMID 9744841
- [Background] Richter KP, Ahluwalia HK, Mosier MC, Nazir N, Ahluwalia JS. A population-based study of cigarette smoking among illicit drug users in the United States. Addiction. 2002 Jul;97(7):861-9. doi: 10.1046/j.1360-0443.2002.00162.x. PMID 12133125
- [Background] Friedmann PD, Jiang L, Richter KP. Cigarette smoking cessation services in outpatient substance abuse treatment programs in the United States. J Subst Abuse Treat. 2008 Mar;34(2):165-72. doi: 10.1016/j.jsat.2007.02.006. Epub 2007 May 23. PMID 17509809
- [Background] Ziedonis DM, Guydish J, Williams J, Steinberg M, Foulds J. Barriers and solutions to addressing tobacco dependence in addiction treatment programs. Alcohol Res Health. 2006;29(3):228-35. PMID 17373414
- [Background] Bobo JK, Davis CM. Recovering staff and smoking in chemical dependency programs in rural Nebraska. J Subst Abuse Treat. 1993 Mar-Apr;10(2):221-7. doi: 10.1016/0740-5472(93)90047-6. PMID 8389899
- [Background] Fuller BE, Guydish J, Tsoh J, Reid MS, Resnick M, Zammarelli L, Ziedonis DM, Sears C, McCarty D. Attitudes toward the integration of smoking cessation treatment into drug abuse clinics. J Subst Abuse Treat. 2007 Jan;32(1):53-60. doi: 10.1016/j.jsat.2006.06.011. Epub 2006 Sep 26. PMID 17175398
- [Background] Myers MG, MacPherson L. Smoking cessation efforts among substance abusing adolescents. Drug Alcohol Depend. 2004 Feb 7;73(2):209-13. doi: 10.1016/j.drugalcdep.2003.09.008. PMID 14725961
- [Background] Hurt RD, Patten CA. Treatment of tobacco dependence in alcoholics. Recent Dev Alcohol. 2003;16:335-59. doi: 10.1007/0-306-47939-7_23. PMID 12638645
- [Background] Satre DD, Gordon NP, Weisner C. Alcohol consumption, medical conditions, and health behavior in older adults. Am J Health Behav. 2007 May-Jun;31(3):238-48. doi: 10.5555/ajhb.2007.31.3.238. PMID 17402864
- [Background] Hser YI, McCarthy WJ, Anglin MD. Tobacco use as a distal predictor of mortality among long-term narcotics addicts. Prev Med. 1994 Jan;23(1):61-9. doi: 10.1006/pmed.1994.1009. PMID 8016035
- [Background] Hurt RD, Offord KP, Croghan IT, Gomez-Dahl L, Kottke TE, Morse RM, Melton LJ 3rd. Mortality following inpatient addictions treatment. Role of tobacco use in a community-based cohort. JAMA. 1996 Apr 10;275(14):1097-103. doi: 10.1001/jama.275.14.1097. PMID 8601929
- [Background] Booth BM, Blow FC, Cook CA, Bunn JY, Fortney JC. Relationship between inpatient alcoholism treatment and longitudinal changes in health care utilization. J Stud Alcohol. 1997 Nov;58(6):625-37. doi: 10.15288/jsa.1997.58.625. PMID 9391923
- [Background] Skog OJ, Duckert F. The development of alcoholics' and heavy drinkers' consumption: a longitudinal study. J Stud Alcohol. 1993 Mar;54(2):178-88. doi: 10.15288/jsa.1993.54.178. PMID 8459712
- [Background] Booth BM, Yates WR, Petty F, Brown K. Patient factors predicting early alcohol-related readmissions for alcoholics: role of alcoholism severity and psychiatric co-morbidity. J Stud Alcohol. 1991 Jan;52(1):37-43. doi: 10.15288/jsa.1991.52.37. PMID 1994121
- [Background] Moos RH, Mertens JR, Brennan PL. Rates and predictors of four-year readmission among late-middle-aged and older substance abuse patients. J Stud Alcohol. 1994 Sep;55(5):561-70. doi: 10.15288/jsa.1994.55.561. PMID 7990466
- [Background] Phibbs CS, Swindle RW, Recine B. Does case mix matter for substance abuse treatment? A comparison of observed and case mix-adjusted readmission rates for inpatient substance abuse treatment in the Department of Veterans Affairs. Health Serv Res. 1997 Feb;31(6):755-71. PMID 9018215
- [Background] Brennan PL, Kagay CR, Geppert JJ, Moos RH. Elderly Medicare inpatients with substance use disorders: characteristics and predictors of hospital readmissions over a four-year interval. J Stud Alcohol. 2000 Nov;61(6):891-5. doi: 10.15288/jsa.2000.61.891. PMID 11188495
- [Background] Ornstein P, Cherepon JA. Demographic variables as predictors of alcoholism treatment outcome. J Stud Alcohol. 1985 Sep;46(5):425-32. doi: 10.15288/jsa.1985.46.425. PMID 2999515
- [Background] Willems S, De Maesschalck S, Deveugele M, Derese A, De Maeseneer J. Socio-economic status of the patient and doctor-patient communication: does it make a difference? Patient Educ Couns. 2005 Feb;56(2):139-46. doi: 10.1016/j.pec.2004.02.011. PMID 15653242
- [Background] Street RL Jr, Gordon HS, Ward MM, Krupat E, Kravitz RL. Patient participation in medical consultations: why some patients are more involved than others. Med Care. 2005 Oct;43(10):960-9. doi: 10.1097/01.mlr.0000178172.40344.70. PMID 16166865
- [Background] Kaplan SH, Gandek B, Greenfield S, Rogers W, Ware JE. Patient and visit characteristics related to physicians' participatory decision-making style. Results from the Medical Outcomes Study. Med Care. 1995 Dec;33(12):1176-87. doi: 10.1097/00005650-199512000-00002. PMID 7500658
- [Background] Nease RF Jr, Brooks WB. Patient desire for information and decision making in health care decisions: the Autonomy Preference Index and the Health Opinion Survey. J Gen Intern Med. 1995 Nov;10(11):593-600. doi: 10.1007/BF02602742. PMID 8583261
- [Background] Cooper LA, Gonzales JJ, Gallo JJ, Rost KM, Meredith LS, Rubenstein LV, Wang NY, Ford DE. The acceptability of treatment for depression among African-American, Hispanic, and white primary care patients. Med Care. 2003 Apr;41(4):479-89. doi: 10.1097/01.MLR.0000053228.58042.E4. PMID 12665712
- [Background] Cooper-Patrick L, Gallo JJ, Powe NR, Steinwachs DM, Eaton WW, Ford DE. Mental health service utilization by African Americans and Whites: the Baltimore Epidemiologic Catchment Area Follow-Up. Med Care. 1999 Oct;37(10):1034-45. doi: 10.1097/00005650-199910000-00007. PMID 10524370
- [Background] Johnson RL, Roter D, Powe NR, Cooper LA. Patient race/ethnicity and quality of patient-physician communication during medical visits. Am J Public Health. 2004 Dec;94(12):2084-90. doi: 10.2105/ajph.94.12.2084. PMID 15569958
- [Background] Street RL Jr. Gender differences in health care provider-patient communication: are they due to style, stereotypes, or accommodation? Patient Educ Couns. 2002 Dec;48(3):201-6. doi: 10.1016/s0738-3991(02)00171-4. PMID 12477604
- [Background] Dawson DA, Grant BF. Gender effects in diagnosing alcohol abuse and dependence. J Clin Psychol. 1993 Mar;49(2):298-307. doi: 10.1002/1097-4679(199303)49:23.0.co;2-z. PMID 8486813
- [Background] Booth BM, McLaughlin YS. Barriers to and need for alcohol services for women in rural populations. Alcohol Clin Exp Res. 2000 Aug;24(8):1267-75. PMID 10968667
- [Background] Roman PM. Biological features of women's alcohol use: a review. Public Health Rep. 1988 Nov-Dec;103(6):628-37. PMID 3141957
- [Background] Hser YI, Anglin MD, McGlothlin W. Sex differences in addict careers. 1. Initiation of use. Am J Drug Alcohol Abuse. 1987;13(1-2):33-57. doi: 10.3109/00952998709001499. PMID 3318399
- [Background] Hser YI, Anglin MD, Booth MW. Sex differences in addict careers. 3. Addiction. Am J Drug Alcohol Abuse. 1987;13(3):231-51. doi: 10.3109/00952998709001512. PMID 3687889
- [Background] Anglin MD, Hser YI, Booth MW. Sex differences in addict careers. 4. Treatment. Am J Drug Alcohol Abuse. 1987;13(3):253-80. doi: 10.3109/00952998709001513. PMID 3687890
- [Background] Marsh JC, Cao D, D'Aunno T. Gender differences in the impact of comprehensive services in substance abuse treatment. J Subst Abuse Treat. 2004 Dec;27(4):289-300. doi: 10.1016/j.jsat.2004.08.004. PMID 15610830
- [Background] Parthasarathy S, Weisner CM. Five-year trajectories of health care utilization and cost in a drug and alcohol treatment sample. Drug Alcohol Depend. 2005 Nov 1;80(2):231-40. doi: 10.1016/j.drugalcdep.2005.04.004. PMID 15916868
- [Background] Clayton RR. Multiple drug use. Epidemiology, correlates, and consequences. Recent Dev Alcohol. 1986;4:7-38. PMID 3486436
- [Background] Kania J, Kofoed L. Drug use by alcoholics in outpatient treatment. Am J Drug Alcohol Abuse. 1984;10(4):529-34. doi: 10.3109/00952998409001490. PMID 6335950
- [Background] Hubbard RL. Treating combined alcohol and drug abuse in community-based programs. Recent Dev Alcohol. 1990;8:273-83. PMID 2185522
- [Background] Weisner C. The merging of alcohol and drug treatment: a policy review. J Public Health Policy. 1992 Spring;13(1):66-80. PMID 1629361
- [Background] Moos RH, Mertens JR, Brennan PL. Patterns of diagnosis and treatment among late-middle-aged and older substance abuse patients. J Stud Alcohol. 1993 Jul;54(4):479-87. doi: 10.15288/jsa.1993.54.479. PMID 8393499
- [Background] Tam TW, Weisner C, Mertens J. Demographic characteristics, life context, and patterns of substance use among alcohol-dependent treatment clients in a health maintenance organization. Alcohol Clin Exp Res. 2000 Dec;24(12):1803-10. PMID 11141039
- [Background] Satre DD, Mertens J, Arean PA, Weisner C. Contrasting outcomes of older versus middle-aged and younger adult chemical dependency patients in a managed care program. J Stud Alcohol. 2003 Jul;64(4):520-30. doi: 10.15288/jsa.2003.64.520. PMID 12921194
- [Background] Liberto JG, Oslin DW, Ruskin PE. Alcoholism in older persons: a review of the literature. Hosp Community Psychiatry. 1992 Oct;43(10):975-84. doi: 10.1176/ps.43.10.975. PMID 1398581
- [Background] Oslin DW. Alcohol use in late life: disability and comorbidity. J Geriatr Psychiatry Neurol. 2000 Fall;13(3):134-40. doi: 10.1177/089198870001300307. PMID 11001136
- [Background] Mertens JR, Weisner CM. Predictors of substance abuse treatment retention among women and men in an HMO. Alcohol Clin Exp Res. 2000 Oct;24(10):1525-33. PMID 11045861
- [Background] Lemke S, Moos RH. Prognosis of older patients in mixed-age alcoholism treatment programs. J Subst Abuse Treat. 2002 Jan;22(1):33-43. doi: 10.1016/s0740-5472(01)00209-4. PMID 11849905
- [Background] Oslin DW, Pettinati H, Volpicelli JR. Alcoholism treatment adherence: older age predicts better adherence and drinking outcomes. Am J Geriatr Psychiatry. 2002 Nov-Dec;10(6):740-7. PMID 12427583
- [Background] Kashner TM, Rodell DE, Ogden SR, Guggenheim FG, Karson CN. Outcomes and costs of two VA inpatient treatment programs for older alcoholic patients. Hosp Community Psychiatry. 1992 Oct;43(10):985-9. doi: 10.1176/ps.43.10.985. PMID 1328022
- [Background] Rice C, Longabaugh R, Beattie M, Noel N. Age group differences in response to treatment for problematic alcohol use. Addiction. 1993 Oct;88(10):1369-75. doi: 10.1111/j.1360-0443.1993.tb02023.x. PMID 8251874
- [Background] Gfroerer J, Penne M, Pemberton M, Folsom R. Substance abuse treatment need among older adults in 2020: the impact of the aging baby-boom cohort. Drug Alcohol Depend. 2003 Mar 1;69(2):127-35. doi: 10.1016/s0376-8716(02)00307-1. PMID 12609694
- [Background] Weisner C, Matzger H, Tam T, Schmidt L. Who goes to alcohol and drug treatment? Understanding utilization within the context of insurance. J Stud Alcohol. 2002 Nov;63(6):673-82. doi: 10.15288/jsa.2002.63.673. PMID 12529067
- [Background] Zeber JE, Copeland LA, Grazier KL. Serious mental illness, aging, and utilization patterns among veterans. Mil Med. 2006 Jul;171(7):619-26. doi: 10.7205/milmed.171.7.619. PMID 16895128
- [Background] Hassan I, McCabe R, Priebe S. Professional-patient communication in the treatment of mental illness: a review. Commun Med. 2007;4(2):141-52. doi: 10.1515/CAM.2007.018. PMID 18052814
- [Background] Holder HD, Blose JO. The reduction of health care costs associated with alcoholism treatment: a 14-year longitudinal study. J Stud Alcohol. 1992 Jul;53(4):293-302. doi: 10.15288/jsa.1992.53.293. PMID 1619923
- [Background] Jerrell JM, Wieduwilt KM, Macey DV. Use and costs of public-sector behavioral health services for african-american and white women. Psychiatr Serv. 2002 Feb;53(2):195-200. doi: 10.1176/appi.ps.53.2.195. PMID 11821551
- [Background] Fleming MF, Mundt MP, French MT, Manwell LB, Stauffacher EA, Barry KL. Benefit-cost analysis of brief physician advice with problem drinkers in primary care settings. Med Care. 2000 Jan;38(1):7-18. doi: 10.1097/00005650-200001000-00003. PMID 10630716
- [Background] Fleming MF, Graham AW. Screening and brief interventions for alcohol use disorders in managed care settings. Recent Dev Alcohol. 2001;15:393-416. doi: 10.1007/978-0-306-47193-3_22. PMID 11449755
- [Background] Fleming MF, Mundt MP, French MT, Manwell LB, Stauffacher EA, Barry KL. Brief physician advice for problem drinkers: long-term efficacy and benefit-cost analysis. Alcohol Clin Exp Res. 2002 Jan;26(1):36-43. PMID 11821652
- [Background] Sterling S, Chi F, Campbell C, Weisner C. Three-year chemical dependency and mental health treatment outcomes among adolescents: the role of continuing care. Alcohol Clin Exp Res. 2009 Aug;33(8):1417-29. doi: 10.1111/j.1530-0277.2009.00972.x. Epub 2009 Apr 30. PMID 19413644
- [Background] Satre DD, Mertens JR, Arean PA, Weisner C. Five-year alcohol and drug treatment outcomes of older adults versus middle-aged and younger adults in a managed care program. Addiction. 2004 Oct;99(10):1286-97. doi: 10.1111/j.1360-0443.2004.00831.x. PMID 15369567
- [Background] Mendelson DN, Schwartz WB. The effects of aging and population growth on health care costs. Health Aff (Millwood). 1993 Spring;12(1):119-25. doi: 10.1377/hlthaff.12.1.119. PMID 8509013
- [Background] Polder JJ, Bonneux L, Meerding WJ, van der Maas PJ. Age-specific increases in health care costs. Eur J Public Health. 2002 Mar;12(1):57-62. doi: 10.1093/eurpub/12.1.57. PMID 11968522
- [Background] Seshamani M, Gray A. Health care expenditures and ageing: an international comparison. Appl Health Econ Health Policy. 2003;2(1):9-16. PMID 14619269
- [Background] Samet JH, Friedmann P, Saitz R. Benefits of linking primary medical care and substance abuse services: patient, provider, and societal perspectives. Arch Intern Med. 2001 Jan 8;161(1):85-91. doi: 10.1001/archinte.161.1.85. PMID 11146702
- [Background] Gordon AJ, Fiellin DA, Friedmann PD, Gourevitch MN, Kraemer KL, Arnsten JH, Saitz R; Society of General Internal Medicine's Substance Abuse Interest Group. Update in addiction medicine for the primary care clinician. J Gen Intern Med. 2008 Dec;23(12):2112-6. doi: 10.1007/s11606-008-0806-7. Epub 2008 Oct 2. No abstract available. PMID 18830761
- [Background] Gordon AJ, Sullivan LE, Alford DP, Arnsten JH, Gourevitch MN, Kertesz SG, Kunins HV, Merrill JO, Samet JH, Fiellin DA. Update in addiction medicine for the generalist. J Gen Intern Med. 2007 Aug;22(8):1190-4. doi: 10.1007/s11606-007-0133-4. Epub 2007 May 10. No abstract available. PMID 17492327
- [Background] Sellers EM, Ciraulo DA, DuPont RL, Griffiths RR, Kosten TR, Romach MK, Woody GE. Alprazolam and benzodiazepine dependence. J Clin Psychiatry. 1993 Oct;54 Suppl:64-75; discussion 76-7. PMID 8262891
- [Derived] Iturralde E, Weisner CM, Adams SR, Chi FW, Ross TB, Cunningham SF, Ghadiali M, Asyyed AH, Satre DD, Campbell CI, Sterling SA. Patterns of Health Care Use 5 Years After an Intervention Linking Patients in Addiction Treatment With a Primary Care Practitioner. JAMA Netw Open. 2022 Nov 1;5(11):e2241338. doi: 10.1001/jamanetworkopen.2022.41338. PMID 36355373
- [Derived] Weisner CM, Chi FW, Lu Y, Ross TB, Wood SB, Hinman A, Pating D, Satre D, Sterling SA. Examination of the Effects of an Intervention Aiming to Link Patients Receiving Addiction Treatment With Health Care: The LINKAGE Clinical Trial. JAMA Psychiatry. 2016 Aug 1;73(8):804-14. doi: 10.1001/jamapsychiatry.2016.0970. PMID 27332703